CLINICAL TRIAL: NCT04835012
Title: Health and Health Care Utilization Effects of Medical Debt Forgiveness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Stanford University (Other); National Opinion Research Center (Other); Abdul Latif Jameel Poverty Action Lab (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Wesley Yin, Associate Professor, University of California, Los Angeles
Other Study IDs: IRB#20-001700
Record Dates: First submitted 2021-03-27; First posted 2021-04-08 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Health Care Utilization; Depression; Anxiety; Subjective Wellbeing
Keywords: Health Care Utilization; Mental Health; Depression; Anxiety; Subjective Wellbeing; Medical Debt
MeSH Terms: conditions — Patient Acceptance of Health Care; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: Subjects in this "treatment" group had their medical debt forgiven by a non-profit charity, RIP Medical Debt. This protocol will administer a survey to measure subjects' health care utilization, mental health, and subjective well-being.
  Interventions: Other: Medical debt forgiveness
- Control: No intervention was given to subjects in this "control" group. This protocol will administer a survey to measure subjects' health care utilization, mental health, and subjective well-being.

INTERVENTIONS:
Other: Medical debt forgiveness — A non-profit charity, RIP Medical Debt, bought and retired medical debt for individuals that were assigned to the treatment group.
  Groups: Treatment

SUMMARY:
The goal of this study is to estimate the direct, causal impact of medical debt on health care utilization, mental health, and wellbeing of patients. The investigators will conduct a survey to measure the impact of the debt forgiveness on health care use, mental health, and wellbeing. The survey will be administered to approximately 17,000 subjects of a recent medical financial intervention. In that prior intervention, a non-profit charity, RIP Medical Debt, purchased and abolished medical debt for a randomly selected about 6,000 (out of the 17,000) individuals. In this current protocol, the investigators will administer the survey, and will compare surveyed outcomes of subjects who received and did not receive the intervention.

DETAILED DESCRIPTION:
This study will estimate the direct, causal impact of medical debt on health care utilization, mental health, and wellbeing of patients. To do so, the investigators will administer a survey to approximately 17,000 subjects of a recent medical financial intervention. In that intervention, a non-profit charity, RIP Medical Debt, purchased and abolished medical debt for a randomly selected about 6,000 (out of the 17,000) study subjects. In this current protocol, the investigators will compare surveyed outcomes of subjects who received and did not receive the medical debt abolishment intervention. Because debt abolishment was randomized, comparing surveyed outcomes of treated and control subjects in the cross-section will allow the study to estimate the causal impact of the medical debt abolishment. The survey will measure the effects of medical debt on three sets of outcomes: (i) health care utilization, as measured by medical care visits, prescription drug utilization and adherence, and unmet need for medical care; (ii) mental health, as measured by validated screens for depression and anxiety; and (iii) subjective wellbeing, as measured by self-reported health, forgone consumption, and financial strain. This study would be the first to provide a direct, causal connection between the rising personal debt associated with U.S. health care and the health outcomes of its recipients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 18 and over who owed medical debt to FFAM, a debt collections agency

Exclusion Criteria:

* Excluded individuals who owed less than $500 in medical debt to FFAM
* Excluded individuals with missing social security numbers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is a probability sample drawn from population of individuals who owe medical debt held by FFAM, a debt collection agency.
Sampling Method: Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
8-item Patient Health Questionnaire (PHQ-8) Depression Scale | An average of 12 months after the intervention.
  Scores on the 8-item Patient Health Questionnaire depression scale range from 0 to 24, with higher scores indicating greater severity of depression.

SECONDARY OUTCOMES:
Received Needed Health Care | An average of 12 months after the intervention.
  Binary response to: "If you needed medical care in the last 12 months, did you get ALL the medical care you needed?" (Health Care Utilization domain)
Received Needed Rx | An average of 12 months after the intervention.
  Binary response to: "If you needed prescription medications in the last 12 months, did you get all the prescription medications you needed?" (Health Care Utilization domain)
7-item Generalized Anxiety Disorder (GAD7) Scale | An average of 12 months after the intervention.
  Scores on the 7-item Generalized Anxiety Disorder Scale range from 0 to 21, with higher scores indicating greater severity of anxiety (Mental Health Domain).
Stress | An average of 12 months after the intervention.
  Binary response to: "Stress means a situation in which a person feels tense, restless, nervous or anxious or is unable to sleep at night because his/her mind is troubled all the time. Do you feel this kind of stress these days?" (Mental Health Domain)
General Health | An average of 12 months after the intervention.
  Response to: "In general, would you say your health is: Excellent, Very Good, Good, Fair, or Poor?" (General Health Domain)
Happiness | An average of 12 months after the intervention.
  Response to: "Taken all together, how would you say things are these days - would you say that you are Very Happy, Pretty Happy, or Not Too Happy?" (Subjective Wellbeing Domain)
Problems paying other bills | An average of 12 months after the intervention.
  Response to: "Besides medical bills, have you had problems paying other types of bills in the past 12 months?" (Financial Stress Domain)
Changes in spending due to medical debt | An average of 12 months after the intervention.
  Indexed response to: "As a result of medical bills have you cut back on spending in the past 12 months on i) basic necessities (like food, heat or housing, or other basic household items), ii) Big-ticket items (like cars, furniture, or appliances); iii) business investments?" (Financial Stress Domain)
Changes in borrowing due to medical debt | An average of 12 months after the intervention.
  Indexed response to: "As a result of medical bills, in the past 12 months, have you i) Increased your credit card debt, or charge card debt? ii) Borrowed money from a payday lender?; iii) Borrowed from friends and family?; iv) Used up all or most of your savings?; v) Increased debt on other lines of credit?" (Financial Stress Domain)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yin, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA IRB, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified and restricted data available to the research community through portals such as the publicly accessible Inter-University Consortium for Political and Social Research (hosted by the University of Michigan). We will preserve the confidentiality of study participants and protect personal health information by stripping the data of personally identifying information and purging it of all personal health information, and any information that is sufficiently fine so that it could identify individuals. We will follow standard protocols, such as converting specific dates to relative dates or date intervals, and aggregating small cells. This will allow us to maximize the data available to researchers while strictly preserving confidentiality and privacy.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: De-identified and confidential IPD will be made available by the on-line publication date of published research.
Access Criteria: Access will be limited to researchers for non-commercial uses. Users will also need to certify that no attempt will be made to re-identify participants from the de-identified data.